CLINICAL TRIAL: NCT06240767
Title: Clinical Study on the Treatment of Advanced Recurrent Tumors With Anticancer Mouse Characteristic Human Neutrophils
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuxi People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WX03-02B0205-072100-62
Record Dates: First submitted 2023-06-12; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-09

CONDITIONS: Solid Tumor, Adult; Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical study of human granulocyte in the treatment of advanced recurrent tumor (Experimental): Experimental: Anticancer mouse characteristic human granulocyte treatment of advanced recurrent tumors.
  A single infusion of human granulocytes with anti-cancer mouse characteristics was performed for 5 consecutive transfusions at a interval of 2±1 day, and the safety and efficacy were clinically observed.
  Interventions: Biological: Granulocyte infusion

INTERVENTIONS:
Biological: Granulocyte infusion — The number of single granulocytes per infusion was 2.0-5.0×10^10, with an interval of 2±1 day and 5 continuous infusions.

SUMMARY:
It is planned to recruit about 100 pathologically confirmed subjects with advanced solid tumors (non-small cell lung cancer, breast cancer, ovarian cancer, stomach cancer, colorectal cancer, pancreatic cancer, mesothelioma, etc.) that have progressed after standard second-line or above treatment such as surgery, chemoradiotherapy, targeted therapy and PD-1 antibody therapy. A single infusion of human granulocytes with anti-cancer mouse characteristics was performed for 5 consecutive transfusions at a interval of 2±1 day, and the safety and efficacy were clinically observed. After the investigator's judgment and discussion with the sponsor, more cycles of treatment can be received after the informed consent is completed until the criteria for stopping treatment are met.

DETAILED DESCRIPTION:
100 cases of advanced cancer with failed chemotherapy or ineffective standard treatment or relief measures were enrolled and clinically observed. Single infusion dose 2.0-5.0 × 1010 granulocytes were continuously infused 5 times every 2 ± 1 day. According to the patient's condition, ensure that the number of subjects with a single tumor is not less than 20.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 ~ 75 years old (inclusive), gender is not limited
2. Malignant tumor confirmed by puncture pathology/postoperative pathology, or PET-CT multi-focal high signal, clinical stage IV
3. Physical status score of 0-2 in ECOG scale
4. Expected survival time ≥3 months
5. Have measurable lesions, calculate the sum of the longest diameter of all target lesions, and report as the baseline sum diameter: the lesions can be accurately measured in at least one direction (record the longest diameter), as long as it conforms to RECIST1.1; If there are multiple lesions, a maximum of 5 lesions (no more than 2 per organ) are required; The efficacy of hematological malignancies such as leukemia can be confirmed by cytology/histology
6. more than 4 weeks have elapsed since previous drug therapy, radiation therapy and surgery; Oral fluorouracil and small molecule targeted drugs required for more than 2 weeks or within 5 half-lives of the drug (whichever is longer)
7. Laboratory tests meet the following criteria: (1) Bone marrow function: absolute count of blood neutrophils (ANC) ≥1*10^9/L, platelets (PLT) ≥75*10^9/L; (2) Liver function: serum total bilirubin (STB), bound bilirubin (CB) ≤ upper limit of normal (ULN) *1.5, alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ULN*2.5 (in the absence of liver metastasis), or ≤ULN*5 (in the presence of liver metastasis); (3) Kidney function: serum creatinine (Cr) ≤ULN*1.5, endogenous creatinine clearance (Ccr) ≥50 mL/min (calculated by Cockcroft-Gault formula)
8. Anti-neutrophil antibody test results are negative
9. The patient volunteered and signed the informed consent

Exclusion Criteria:

* 1: Uncontrolled or severe cardiovascular disease, diabetes, major heart disease, such as arrhythmia within 30 days, congestive heart failure, or severe coronary artery disease

  2: HIV infection, no recent (within 30 days) use of immunosuppressive drugs other than steroids

  3: Pregnant and lactating women

  4: Previous history of stem cell and organ transplantation

  5: Patients who have been using or are using immunosuppressants for a long time

  6: Symptomatic brain metastases are not controlled

  7: People who are known to be severely allergic to granulocyte infusion (or test positive for anti-neutrophil antibodies)

  8: People with coagulation disorders

  9: Mental disorders are not under control

  10: Patients with severe autoimmune diseases

  11: Cases deemed unsuitable for inclusion by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy evaluation | 6 months after treatment
  Target lesions were assessed according to RECIST1.1 criteria. All other lesions, including small lesions (lesions with a maximum diameter of less than 20mm measured by conventional methods or less than 10mm measured by spiral CT scanning, or less than 15mm measured when the CT layer thickness is 5mm) and true unmeasurable lesions are not required to be measured, described as "with" or "without".

CONTACTS AND LOCATIONS:
Locations (1):
- Wuxi People's Hospital, Wuxi, Jiangsu, China